CLINICAL TRIAL: NCT04114149
Title: Effective Postoperative Pain Relief After Laparoscopic Cholecystectomy With TENS (Transcutaneous Electrical Nerve Stimulation) Treatment for First Line of Treatment Compared to Conventional Treatment With Opioids
Brief Title: Effective Postoperative Pain Relief After Laparoscopic Cholecystectomy With TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUREG-832941/ 249891
Record Dates: First submitted 2019-04-23; First posted 2019-10-03 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative
Keywords: Pain; Transcutaneous Electric Nerve Stimulation; Analgesics, Opioid
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Transcutaneous Electric Nerve Stimulation; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TENS (transcutaneous electrical nerve stimulation) (Active Comparator): High frequency, high intensity TENS treatment. Patients who report postoperative pain intensity according to NRS (numeric rating scale) ≥ 3 during the time spent in post-anesthesia care unit.
  Interventions: Device: TENS (transcutaneous electrical nerve stimulation)
- Conventional treatment with iv opioid (Active Comparator): Patients who report postoperative pain intensity according to NRS (numeric rating scale) ≥ 3 during the time spent in post-anesthesia care unit.
  Interventions: Drug: iv opioid
- Control (No Intervention): Patients who report postoperative pain intensity according to NRS (numeric rating scale) < 3 during the time spent in post-anesthesia care unit.

INTERVENTIONS:
Device: TENS (transcutaneous electrical nerve stimulation) — TENS as first line of treatment. If insufficient pain relief, i.e. postoperative pain intensity according to NRS (numeric rating scale) ≥ 3 after two treatment sessions à 1 minute, the patient receives conventional treatment with iv opioids.
  Arms: TENS (transcutaneous electrical nerve stimulation)
Drug: iv opioid — Conventional treatment with iv opioid if postoperative pain intensity according to NRS (numeric rating scale) ≥ 3.
  Arms: Conventional treatment with iv opioid

SUMMARY:
The study evaluates the effect of TENS (transcutaneous electrical nerve stimulation) treatment for first line of treatment compared with conventional treatment with opioids on pain relief and time spent time in the post-anesthesia care unit after laparoscopic cholecystectomy. Half of the patients are randomized to TENS as first line of treatment and the second half is randomized to conventional opioid treatment. Patients who does not report postoperative pain which requires treatment are used as controls.

DETAILED DESCRIPTION:
Postoperative pain is often a problem after laparoscopic cholecystectomy. Conventional treatment with intravenous (iv) opioids often offers satisfactory pain relief. However, opioids have negative side effects, such as sedation, nausea, and respiratory depression. Some of these side effects require monitoring of the patient, resulting in longer duration of stay in the post-anesthesia care unit (PACU) after surgery. Transcutaneous electrical nerve stimulation (TENS) has been used to provide pain relief in various postoperative pain conditions. Previous studies from the investigator's center indicate that TENS treatment for postoperative pain after gynecological surgery results in shorter time in the PACU.

Previous studies indicate that patients reporting pain intensity associated with venous cannulation to > 2 VAS (visual analog scale) units have higher risk of postoperative pain in the PACU. The aim of the study is to compare time spent in the PACU and to compare the postoperative pain relieving effect of high frequency, high intensity TENS as first line of treatment with conventional treatment with iv opioids in patients undergoing laparoscopic cholecystectomy. Furthermore, the study evaluates if postoperative opioid consumption can be reduced by using TENS as first line of treatment. In addition, the study tests if pain intensity associated with venous cannulation can be used to predict occurrence of postoperative pain.

Addmendment after study registration:

166 participants were randomized in the RCT part of the study. In the observational part of the study (investigating if pain intensity associated with venous cannulation can be used to predict occurrence of postoperative pain) 258 participants were included. The ethical application (approval number 954-18) covers both parts of the study (i.e. RCT and observaltional study).

ELIGIBILITY:
Inclusion Criteria:

For randomized patients:

• Patients who reports postoperative pain intensity ≥ 3 according to numeric rating scale during the stay in the post-anesthesia care unit after laparoscopic cholecystectomy.

For controls:

• Patients who reports postoperative pain intensity <3 according to numeric rating scale during the stay in the post-anesthesia care unit after laparoscopic cholecystectomy

Exclusion Criteria:

(for all patients)

* Patients who do not want to participate in the study
* Patients younger than 18 years
* Inadequate knowledge of the Swedish language
* Patients with pacemaker or internal cardioverter defibrillator
* Patients who preoperatively report continuous opioid consumption
* Patients with chronic pain conditions
* Patients with impaired sensibility over the dermatomes that are to be treated with TENS
* Alcohol or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Time spent in post-anesthesia care unit | Up to 24 hours after surgery
  Time spent in post-anesthesia care unit in minutes after laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
PAIN NRS | Continuous assesment during the time spent in post-anesthesia care unit, up to 24 hours after surgery
  Pain intensity according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to postoperative pain.

OTHER OUTCOMES:
Time to pain relief | From debut of pain to pain relief, as defined above, during the time spent in post-anesthesia care unit, up to 24 hours after surgery
  Time (in minutes) from debut of postoperative pain intensity ≥ 3 according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to postoperative pain, to pain relief defined as pain intensity according to numeric rating scale <3.
Consumption of analgesics | Assesment during the time spent in post-anesthesia care unit, up to 24 hours after surgery
  Consumption of analgesics during the time spent in post-anesthesia care unit
Patient treatment satisfaction according to NRS | Assesment at end of post-anesthesia care unit stay, up to 24 hours after surgery
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 1 day after surgery
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 7 days after surgery
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Time spent in hospital | From arrival at the post-anesthesia care unit to end of hospital stay, an average of 1-2 days
  Time spent in hospital in hours in relation to undergoing laparoscopic cholecystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Paulin Andréll, MD, PhD, Principal Investigator — Göteborgs Universitet/Västra Götalands Regionen
Locations (1):
- Frölunda Specialistsjukhus, Gothenburg, Västra Götalands Regionen, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelini E, Josefsson C, Ogren C, Andrell P, Wolf A, Ringdal M. Patients experiences of TENS as a postoperative pain relief method in the post-anesthesia care unit after laparoscopic cholecystectomy: a qualitative study. BMC Anesthesiol. 2025 Jan 9;25(1):18. doi: 10.1186/s12871-024-02872-4. PMID 39789467